CLINICAL TRIAL: NCT05660941
Title: An Open-label, Single-centre, Randomised, Two-period, Cross-over Study to Assess the Efficacy and Safety of Automated Closed-loop Glucose Control in Adults With Type 1 Diabetes Comparing Ultra-fast Acting Insulin Lispro With Insulin Lispro
Brief Title: Automated Fully Closed-Loop Insulin Delivery in Type 1 Diabetes With Ultra-Rapid Lispro (ACOLYTE Study)
Acronym: ACOLYTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B01661
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Type 1; Closed Loop; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrarapid-acting Lispro (Experimental): ultrarapid-acting lispro delivered by hybrid closed loop system.
  Interventions: Drug: Lispro
- Insulin Lispro (Active Comparator): Insulin lispro delivered by hybrid closed loop system.
  Interventions: Drug: Lispro

INTERVENTIONS:
Drug: Lispro — Ultra rapid Lispro
  Other Names: Lyumjev
  Arms: Ultrarapid-acting Lispro
Drug: Lispro — Conventional Lispro
  Other Names: Humalog
  Arms: Insulin Lispro

SUMMARY:
The main objective of the study is to determine whether fully closed-loop insulin delivery using ultra-rapid acting insulin lispro will improve glucose control compared to standard lispro under conditions mimicking missed meal bolus. Ultra-rapid acting lispro (Lyumjev) is a novel formulation of insulin lispro in which two additional excipients (citrate and trepostinil) have been added, resulting in accelerated initial absorption and more than double the glucose lowering effect in the first 30 minutes after subcutaneous administration using insulin pump. To date, no randomised controlled trial involving fully closed-loop in type 1 diabetes has been performed to evaluate the benefit of Lyumjev over standard lispro.

This is an open-label, single-centre, two-period, randomised, crossover study. The study involves two 12-hour in-patient stays at the clinical research facility during which glucose levels will be controlled by the Cambridge closed-loop system with either Lyumjev or standard lispro. Up to 26 adults with type 1 diabetes treated with insulin pump will be recruited at Manchester Royal Infirmary, aiming for 19 completed participants.

During the study days, closed-loop will automatically modulate insulin infusion rate based on real-time glucose sensor measurements. Participants will receive standardised meals with no meal bolus for the lunch time meal during each study day. Primary outcome is the time spent in sensor glucose range (3.9-10.0mmol/l) between 11:00 - 17:00 hrs. Secondary outcomes are the time spent with glucose levels above and below target, and other sensor-based metrics. Safety evaluation comprises assessment of the frequency of hypo and hyperglycaemic episodes.

DETAILED DESCRIPTION:
Study Design An open-label, single-centre, randomised, 2-period cross-over study, in adults (18 years and older) with type 1 diabetes on insulin pump treatment.

It is expected that up to 26 adults with type 1 diabetes will be recruited, aiming for 19 completed participants. The study flow chart is outlined in Figure 2.

Study Subjects Study Population This is a single centre study and recruitment will take place at the Manchester Diabetes Centre, Manchester Royal Infirmary, Manchester University NHS Foundation Trust. Up to a total of 26 adults aged 18 years and older with type 1 diabetes on insulin pump therapy will be recruited aiming for 19 completed participants. Potential participants will be identified by their treating clinicians and invited to contact the research team. They will be sent the study information leaflets and an invitation to join the study by the research team.

Randomisation Eligible subjects will be randomised by the clinical researcher up to 14 days prior to first in-patient stay using Sealed Envelope randomisation software to undertake closed-loop studies in one of two possible random sequences; ultrarapid-acting lispro followed by insulin lispro, or insulin lispro followed by ultrarapid-acting insulin lispro.

Study Schedule Overview The study will be co-ordinated from the Manchester Diabetes Centre, Manchester Royal Infirmary, Manchester. The study will consist of five Visits including two 9-hour stays at the MCRF, Manchester Royal Infirmary, Manchester. Visits 1 and 2 may be combined. Tables 1 and 2 summarise the study visits.

Recruitment Visit and Baseline Assessment (Visit 1)

Once the subjects have agreed to participate in the study, they will be invited for the recruitment visit, when the following activities will be performed by the research team:

* Written informed consent
* Checking inclusion and exclusion criteria
* Medical (diabetes) history
* Body weight and height measurement; calculation of BMI
* Record of current insulin therapy
* Serum pregnancy test (females of child-bearing potential) Baseline Blood Sampling During Visit 1 consented participants will undergo a baseline evaluation where blood samples for HbA1c and serum beta HCG (pregnancy test) in females of child-bearing potential will be collected. Less than 15 ml of whole blood will be taken from each participant. In the event the laboratory HbA1c returns below 48 mmol/mol or above 86 mmol/mol the participant will be withdrawn.

Training Session on Continuous Glucose Monitoring (Visit 2) This session will cover key aspects of the study CGM and attention will be paid to the following areas. This visit could be combined with visit 1.

* Insertion and initiation of sensor session
* Sensor calibrations
* Use of CGM data to optimise treatment

Written easy to use guidelines for the operation of CGM device will be provided. This session will be conducted by a professional pump educator / study nurse and possibly a member of the study team. Competency on the use of CGM will be assessed and additional training will be provided if deemed necessary by the Competency Assessment Form.

Visit 3 - Optimisation During Visit 3, after a 2 to 3 weeks' run-in period, glucose control will be optimised, if required, by the study team with special focus on insulin to carbohydrate ratios.

Manchester Diabetes Centre is the largest insulin pump centre in UK. We expect most of the participants in the study to be already well optimised. However, we will ensure this further by reviewing insulin, glucose and carbohydrate data during the two-week run-in period. Particular attention will be on the insulin carbohydrate ratio to see whether it is over aggressive. If the insulin to carb ratio is over aggressive this could potentially reduce the difference between Lispro and Lyumjev during the study. Participants whose glucose levels drops (those who develop hypoglycaemia within 2 to 3 hours of meal bolus) carb ratio will be adjusted to avoid this drop. Participants will also be randomised at visit 3.

Visit 4 will follow within 2 weeks of Visit 3. Participants will be advised to avoid strenuous exercise 24 hours prior to each in-patient stay to avoid any bias arising from changes in insulin sensitivity.

Activities during 9-hour in-patient stay (Visits 4 and 5, Figure 3) There will be two in-patient study days, performed within 1-6 weeks of each other. On each Study Day, participants will arrive at the study centre at approximately 08.30 and will be discharged by 18.00 the same day.

Participants will be advised to insert a new CGM sensor 48 hours before the planned admission. A new insulin infusion cannula will be inserted on admission to the clinical research facility. In addition, participant will be advised to change their usual insulin to the corresponding study visit insulin formulation, 24 hours prior to admission. (For example; if the participant is on insulin lispro, this will be changed to ultra rapid-acting lispro 24-hour prior to the admission for closed loop with ultrarapid-acting lispro and vice versa.) Participants will be requested to fast from 12 midnight prior to admission (carbohydrate-free liquids are allowed). Participants will be requested to check their glucose between 05:00 and 07:00. If the glucose level is, or anticipated to be, < 4 mmol/l during this period, additional carbohydrate can be taken to aim for arrival glucose between 4 and 10 mmols. Correction insulin doses may be given if arrival glucose is anticipated to be above range (>10 mmol/l). Study visits may be rescheduled if participants develop significant hypoglycaemia (<3.0 mmol) or significant hyperglycaemia (glucose >20 mmol/l and/or ketones >0.6 mmol/l) 6 hours prior to or on arrival. On arrival, participant's usual insulin pump will be changed to study insulin pump. Closed-loop with either ultrarapid-acting lispro or insulin lispro will commence between 09:00 and 17:00 hours.

A 60g meal will be served at 11:00 with no meal bolus to mimic a missed meal bolus.

The study will end at 17.00. Patients will be switched back to their usual insulin pump therapy at the end of the study. Standard operating procedures will be in place for treatment of hypo and hyperglycaemia. Figure 3 summarises activities during the 9 hour in-patient stay.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18 years or older 2. Type 1 diabetes, as defined by WHO, for at least 1 year or confirmed C-peptide negative 3. An insulin pump user for at least 3 months 4. Treated with any of the rapid acting insulin analogues (Insulin aspart, faster acting aspart, insulin lispro, ultra-rapid acting lispro or insulin glulisine) 5. Willing to adhere to study procedures 6. HbA1c ≥ 6.5% (48 mmol/mol) and ≤ 10 % (86mmol/mol) based on analysis from local laboratory or equivalent within 36 months of enrolment or estimated HbA1c (GMI) based on sensor glucose data 7. Literate in English

Exclusion Criteria:

1. Non-type 1 diabetes mellitus including those secondary to chronic disease
2. Any other physical or psychological disease likely to interfere with the normal conduct of the study
3. Untreated celiac disease or hypothyroidism
4. Clinically significant nephropathy, neuropathy or proliferative retinopathy as judged by the investigator
5. Total daily insulin dose equal or more than 2 U/kg/day
6. Total daily insulin dose < 10 U/day
7. Pregnancy, planned pregnancy, or breast feeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Time in range | 6 hours
  The primary outcome is time spent in the target glucose range (3.9 to 10.0 mmol/l) based on sensor glucose levels, between the hours of 11:00 and 17:00 hours, during inpatient stay

SECONDARY OUTCOMES:
Area under curve | 4 hours
  • Incremental area above the curve of sensor glucose level during the first 4 hours after the meal.
Time below target | 6 Hours
  Time spent below target glucose (<3.9mmol/l)
Time above target | 6 Hours
  Time spent abovetarget glucose (10.0mmol/l)
Mean glucose and glycaemic variability | 6 hours
  Average, coefficient of variation and standard deviation glucose levels
Insulin dose | 6 hours
  Total, basal and bolus insulin dose
Time above and below significant sensor glucose levels | 6 hours
  The time with sensor glucose levels < 3.5 mmol/l, 3.0 and <2.8 mmol/l and the time with sensor glucose levels in the significant hyperglycaemia (glucose levels > 16.7 mmol/l)

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided